CLINICAL TRIAL: NCT06623357
Title: Pilot Test of Caregiver Training Protocol for Brachial Plexus Birth Injury
Acronym: CTP-BPBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Towson University (Other)
Responsible Party: Principal Investigator, Matthew Elrick, Pediatric Neurologist, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00450720
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Brachial Plexus Birth Palsy; Erbs Palsy
Keywords: Brachial Plexus Birth Injury; Brachial Plexus; Passive Range of Motion; Caregiver Education; Caregiver Training; Contracture
MeSH Terms: conditions — Brachial Plexus Neuropathies; Contracture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Pilot Protocol (Experimental): Participants in Group A will receive training in PROM techniques via a visual handout with pictures and written instructions and video recording using the caregiver's cell phone/tablet of the trainer and/or caregiver performing PROM on the infant. Participants in Group A will also receive supplemental training including a step-by-step checklist for each of the shoulder stretches that are recommended and will be instructed to refer to the checklist each time they perform PROM at home. Participants will be observed performing PROM at their initial visit where training occurs and at their infants' next follow-up visit. The standardized checklist will be used to assess efficacy of caregivers' demonstrated PROM including assessment of positioning, hand placement, and number of cues needed to facilitate accuracy; specific feedback will be given as needed.
  Interventions: Other: Pilot Training Protocol
- Group B - Standard Protocol (Active Comparator): Participants in Group B will receive training in PROM techniques via the same visual handout with pictures and written instructions provided to Group A as well as video recording using the caregiver's cell phone/tablet of the trainer and/or caregiver performing PROM on the infant.
  Interventions: Other: Standard Training Protocol

INTERVENTIONS:
Other: Pilot Training Protocol — The pilot training protocol uses principles based on evidence-based research on factors that support caregiver learning of and adherence to home-therapy techniques/recommendations.
  Arms: Group A - Pilot Protocol
Other: Standard Training Protocol — The standard training protocol uses the caregiver training methods that are currently used in our clinics.
  Arms: Group B - Standard Protocol

SUMMARY:
The brachial plexus is a network of nerves that exit the spinal cord from the C5-T1 nerve roots and provide all motor and sensory function to the arm from the shoulder to the fingers. Injury to the brachial plexus due to traction forces during labor and/or delivery causing the nerves to stretch or tear occurs in 0.9 out of 1000 live births. As many as 30% of infants with brachial plexus birth injury (BPBI) have paralysis or weakness in one arm resulting in lifelong impairment in arm function with joint contractures, the shortening of tendons, ligaments and muscles, leading to reduced range of motion (ROM), being a common complication and major source of disability. A primary goal of early management of BPBI is to use passive range of motion (PROM) (stretching) to improve and/or maintaining shoulder ROM due to the known risk of shoulder contracture within the first year of life. Infants who develop contractures face challenges in overall sensory-motor development and are less able to participate in meaningful occupations and activities of daily living due to limited upper extremity ROM. They are also at risk for subsequent surgeries throughout their lives. Occupational therapy practitioners (OTPs) and physicians who specialize in treating infants with BPBI recommend caregivers to perform PROM at every diaper change, which is every 1-3 hours in the first months of life, and every 4-6 hours by age one. A survey study by one of the investigators on this proposed project found that 85% of OTPs who specialize in BPBI make this recommendation for performing PROM at every diaper change; however, there is no research to support this frequency to prevent or decrease contractures. Clinical observations suggest that infants who receive consistent daily PROM seem to avoid development of shoulder contractures while those who receive no or infrequent PROM seem to develop early and significant contractures. In a retrospective pilot study we found that children whose parents consistently performed PROM two times daily starting before age two months were less likely to develop shoulder contractures than children whose parents were inconsistent in performing PROM. These findings, along with our clinical observations suggest that frequency of PROM might be less important than consistency. In order to assess the efficacy of different levels of frequency (e.g., at every diaper change vs. two times per day), it is imperative to identify methods that support caregivers in performing PROM every day. Therefore, the proposed study will pilot a caregiver training method which, if successful in facilitating daily adherence, will be used as part of a larger planned study that will compare differences in recommended frequencies of stretching.

In a survey study and scoping literature review performed by one of the co-investigators on this project, caregiver adherence to home therapy recommendations was found to be facilitated by confidence in the training they received and by their confidence in ability to carry-out recommendations; lack of confidence in performing the home therapy recommendations was found to be a common barrier. Therefore, the objective of the proposed work is to assess the efficacy of a pilot training protocol for caregivers of infants with BPBI. Our central hypothesis is that the pilot training protocol will improve caregiver efficacy and increase their confidence in performing the recommended PROM/stretching procedure, thus facilitating adherence which we hope to later demonstrate will decrease the risk of shoulder contracture in infants with BPBI. The significance of this work is that it will evaluate and provide evidence for the use of the pilot training protocol so that this training protocol can later be used in a larger study on the efficacy of different frequencies of PROM to reduce the development of shoulder contracture in infants with BPBI, and thus contribute to developing evidenced-based standards of care for this population.

The objectives of this clinical trial are to:

1. determine whether caregivers who receive a pilot training protocol for performing PROM demonstrate improved efficacy in performing PROM compared to caregivers who receive standard training
2. determine whether caregivers who receive a pilot training protocol for performing PROM demonstrate improved self-confidence in performing PROM compared to caregivers who receive standard training
3. determine whether caregivers who receive a pilot training protocol for performing PROM report better daily adherence to daily PROM compared to caregivers who receive standard training

DETAILED DESCRIPTION:
The proposed project is a prospective multi-site randomized trial. Participants will be recruited from two JHMI affiliated multidisciplinary brachial plexus clinics: Kennedy Krieger Institute (KKI) and Johns Hopkins All Children's Hospital (ACH) in St. Petersburg, Florida. Both clinics are led by investigator, Dr. Allan Belzberg; the PI Dr. Matt Elrick is the neurologist at KKI's clinic. Co-investigator Jennifer Wingrat is the senior occupational therapist at KKI's clinic and Lisa Tetreault is Clinic Coordinator at ACH. Both clinics meet monthly with an average of two new patients and up to 10 follow-up patients per clinic each month. Caregivers of all new patients up to 6 months of age will be eligible to enroll in the study, with enrollment continuing until we reach 20 participants, which we anticipate will occur within 12 months. The sample size of 20 was chosen due to the feasibility of recruiting participants based on the typical demographics of the two clinics from which participants are being recruited; because this is a pilot study, the sample size should be sufficient to provide preliminary data. As recruitment will occur on a rolling basis, no interim data analyses are planned.

When a new patient is scheduled at either of the JHMI brachial plexus clinics, J. Wingrat or Lisa Tetreault will contact the primary caregiver via phone or email to describe the study and to obtain verbal consent; virtual meeting via FaceTime or Zoom will be offered to provide information about the study if desired. Signed consent will be obtained when the caregiver brings their child to their first scheduled clinic appointment. Enrolled caregivers will be randomly assigned to one of two equally sized intervention groups. Group A will be instructed in the pilot PROM training protocol and Group B will receive standard training. Caregiver instruction in PROM provided by the occupational therapist is part of routine care for all infants with a BPBI seen in the clinic.

Per routine clinic protocol, all caregivers will receive training in PROM techniques via a visual handout with pictures and written instructions and video recording using the caregiver's cell phone/tablet of the clinic-therapist and/or caregiver performing PROM on the infant. The caregivers of infants in group A, the pilot training group, will receive supplemental training including a step-by-step checklist for each of the shoulder stretches that are recommended. Caregivers in Group A will be instructed to refer to the checklist each time they perform PROM at home. J. Wingrat and or L. Tetreault will provide the training at each participant's first clinic visit.

Caregivers will be observed performing PROM at their initial visit where training occurs and at their infants' next follow-up visit. The standardized checklist will be used to assess the efficacy of caregivers' demonstrated PROM which includes assessment of positioning, hand placement, and number of cues needed to facilitate accuracy. Caregivers in Group A (the pilot group) will receive specific feedback based on the checklist. Caregivers' perception of self-confidence will be measured using a survey after initial training is provided and at their infant's next follow-up visit; the follow-up survey will also ask caregivers to self-report how frequently they performed PROM. Per routine clinic protocol, active range of motion will be assessed and documented for all infants using the Active Movement Scale at the initial visit and again at the follow-up visit. All data will be entered into a de-identified data record form and stored in a password-protected file in the JHMI SAFE Desktop application. The study will be stopped early if the researchers become aware of new evidenced-based data on a caregiver training protocol for PROM for infants with BPBI.

Study duration will be up to three years with rolling enrollment of caregivers of newly referred infants as they are referred to either of the two clinics. Caregivers of infants between birth and 6 months of age will be eligible for enrollment and will remain enrolled until their child's first follow-up visit, resulting in two total study visits per participant.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver, age 18+ of an infant age 6 months or younger with a confirmed BPBI determined by the brachial plexus clinic team at an infant's first visit

Exclusion Criteria:

* Caregiver of an infant older than 6 months of age scheduled at the brachial clinic Caregiver of an infant scheduled at the brachial plexus clinic with a diagnosis other than BPBI and/or co-morbidity known to cause joint contractures
* Caregiver of infant with BPBI who requires surgery prior to nine months of age
* Caregiver who does not speak English unless a JHMI interpreter is present at the clinic visit, at which point a short form consent will be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Caregiver Efficacy and Self-Confidence | From enrollment at initial visit to first follow up visit within 1-6 months
  Caregiver efficacy and self-confidence will be measured using surveys completed after their initial training and again at their child's follow-up clinic visit. Average scores will be computed for all surveys and independent t-tests will compare differences in mean scores for caregiver efficacy and self-confidence for the group receiving the pilot training and the group receiving the standard training.

SECONDARY OUTCOMES:
Caregiver self-report of frequency of daily PROM (stretching) | From enrollment until first follow-up visit at 1-6 months
  Independent t-tests will compare number of times per day PROM was performed as reported by participants in each group. 2. Correlation coefficients will be computed to assess relationship between caregiver self-reported efficacy and number of times per day that PROM was performed, and 2) care-giver self-reported confidence and number of times per day that PROM was performed

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Elrick, MD, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (2):
- United States (2):
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Kennedy Krieger Institute, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
All study outcomes will be reported in the aggregate

REFERENCES:
- [Background] Smith BW, Daunter AK, Yang LJ, Wilson TJ. An Update on the Management of Neonatal Brachial Plexus Palsy-Replacing Old Paradigms: A Review. JAMA Pediatr. 2018 Jun 1;172(6):585-591. doi: 10.1001/jamapediatrics.2018.0124. PMID 29710183
- [Background] Wingrat J, Price C, Wright T. Facilitators of and Barriers to Caregiver Adherence to Home Therapy Recommendations for Infants and Children With Neuromotor and Neuromuscular Diagnoses: A Scoping Review. Am J Occup Ther. 2024 Sep 1;78(5):7805205070. doi: 10.5014/ajot.2024.050567. PMID 39083636
- [Background] Wingrat J, Elrick MJ. Frequency, facilitators, and barriers for range of motion to prevent shoulder contracture in brachial plexus birth injury: A pilot study. J Pediatr Rehabil Med. 2023;16(2):331-336. doi: 10.3233/PRM-220090. PMID 37005904
- [Background] DeFrancesco CJ, Shah DK, Rogers BH, Shah AS. The Epidemiology of Brachial Plexus Birth Palsy in the United States: Declining Incidence and Evolving Risk Factors. J Pediatr Orthop. 2019 Feb;39(2):e134-e140. doi: 10.1097/BPO.0000000000001089. PMID 29016426